CLINICAL TRIAL: NCT01129518
Title: An Open Label Randomised Controlled Study to Evaluate the Induction of Immune Memory Following Infant Vaccination With a Glycoconjugate Neisseria Meningitidis Serogroup C Vaccine and to Assess the Immunological Impact of Administering Routine Infant Immunisations in Consistent Versus Alternating Limbs
Brief Title: Can we Reduce the Number of Vaccine Injections for Children?
Acronym: MALTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008_06
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Invasive Meningococcal Disease
Keywords: meningococcal serogroup C; vaccine; conjugate
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Two Dose MenC Group (Experimental): Two doses of MenC-CRM197 priming at 3 and 4 months of age.
  Interventions: Biological: Glyco-conjugate Neisseria meningitidis serogroup C (MenC) vaccine; Biological: Routine schedule immunisations except monovalent MenC vaccine
- Single Dose MenC-CRM197 Group (Experimental): One dose of MenC-CRM197 priming at 3 months of age.
  Interventions: Biological: Glyco-conjugate Neisseria meningitidis serogroup C (MenC) vaccine; Biological: Routine schedule immunisations except monovalent MenC vaccine
- Single Dose MenC-TT Group (Experimental): Single dose MenC-TT priming at 3 months of age
  Interventions: Biological: Glyco-conjugate Neisseria meningitidis serogroup C (MenC) vaccine; Biological: Routine schedule immunisations except monovalent MenC vaccine
- Control Group (Experimental): Zero dose MenC priming
  Interventions: Biological: Routine schedule immunisations except monovalent MenC vaccine

INTERVENTIONS:
Biological: Glyco-conjugate Neisseria meningitidis serogroup C (MenC) vaccine — In order to ensure proper intramuscular injection of the study vaccines, a 23G (0.5mm in diameter) needle of at least 1 inch (2.54 cm) length will be used. All vaccines will be administered intramuscularly.
  Then MenC vaccine will administered either once (at 3 months) or twice (at 3 and 4 months) depending on treatment group to either the thigh, deltoid or a combination of the two.
  Arms: Single Dose MenC-CRM197 Group; Single Dose MenC-TT Group; Two Dose MenC Group
Biological: Routine schedule immunisations except monovalent MenC vaccine — Routine schedule immunisations will be given according to NHS guidelines.

SUMMARY:
This open label randomised controlled study will evaluate the induction of immunity following varying schedules of vaccination with glyco-conjugate Neisseria meningitidis serogroup C (MenC) vaccines in infancy. 498 infants will be enrolled in this multi-centre trial. Participants will receive either 0, 1, or 2 priming doses of a MenC-CRM197 conjugate vaccine or 1 priming dose of a MenC-TT conjugate vaccine in the first year of life, with all groups receiving a dose of a combination Hib-MenC-TT vaccine at 12 months, as well as all other concurrent routine vaccinations. All groups will also be further divided into 2 groups to receive their routine vaccines in either consistent or alternating limbs to assess the immune response to the concurrent infant routine immunisations administered in consistent versus alternating limbs. Immune responses will be assessed at 5, 12, 12months +6 days, 13 and 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infants aged 6-12 weeks at the time of the first vaccination and who were born between 37 and 42 weeks of gestation
* Infants who are known to be free from medical problems as determined by a medical history and clinical examination
* Parents or guardians who are willing for their child to participate and who would be expected to comply with the requirements of the protocol
* Parents/guardians who have given informed consent for their child's participation in the study

Exclusion Criteria:

* History of invasive meningococcal C disease
* Previous vaccination against meningococcal serogroup C disease
* Planned administration/administration of vaccines, since birth, other than the study vaccines (with the exception of oral rotavirus vaccine, Hepatitis B vaccine and BCG).
* Receipt of investigational vaccines/drugs, other than the vaccines used in the study, within 30 days prior to receiving the first dose of the vaccines or their planned use during the study period
* Confirmed or suspected immunosuppressive or immunodeficient conditions, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* Receipt of more than 2 weeks of immunosuppressants or immune modifying drugs, (e.g. prednisolone >0.5mg/kg/day)
* History of allergy to any component of the vaccines.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures
* Acute disease at the time of recruitment as defined by the presence of a moderate or severe illness with or without fever (with the exception of minor illnesses such as diarrhoea, mild upper respiratory infection without fever). In such situations enrolment should be postponed until the participant has recovered.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period
* Parents who plan to move out of the geographical area where the study would be conducted.

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 404 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Geometric mean titres (GMTs) of meningococcal serogroup C (MenC) specific serum bactericidal antibodies, using rabbit complement (rSBA) | 1 month after a 12 month dose of Hib-MenC vaccine
  To demonstrate non-inferiority of the geometric mean titres (GMTs) of meningococcal serogroup C (MenC) specific serum bactericidal antibodies, using rabbit complement (rSBA), 1 month after a 12 month dose of Hib-MenC vaccine in children receiving a single dose of MenC-CRM197vaccine at 3 months of age (single dose priming) compared with those receiving 2 doses at 3 and 4 months of age (2 dose priming).

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Vaccine Group, Oxford, United Kingdom

REFERENCES:
- [Derived] Pace D, Khatami A, Attard-Montalto S, Voysey M, Finn A, Faust SN, Heath PT, Borrow R, Snape MD, Pollard AJ. Use of a booster dose of capsular group C meningococcal glycoconjugate vaccine to demonstrate immunologic memory in children primed with one or two vaccine doses in infancy. Vaccine. 2016 Dec 7;34(50):6350-6357. doi: 10.1016/j.vaccine.2016.10.038. Epub 2016 Oct 28. PMID 28029540
- [Derived] Pace D, Khatami A, McKenna J, Campbell D, Attard-Montalto S, Birks J, Voysey M, White C, Finn A, Macloed E, Faust SN, Kent AL, Heath PT, Borrow R, Snape MD, Pollard AJ. Immunogenicity of reduced dose priming schedules of serogroup C meningococcal conjugate vaccine followed by booster at 12 months in infants: open label randomised controlled trial. BMJ. 2015 Apr 1;350:h1554. doi: 10.1136/bmj.h1554. PMID 25832102
- [Derived] Iro MA, Khatami A, Marshall AS, Pace D, Voysey M, McKenna J, Campbell D, Attard-Montalto S, Finn A, White C, Faust SN, Kent A, Heath PT, MacLeod E, Stanford E, Findlow H, Almond R, Bai X, Borrow R, Snape MD, Pollard AJ. Immunological effect of administration of sequential doses of Haemophilus influenzae type b and pneumococcal conjugate vaccines in the same versus alternating limbs in the routine infant immunisation schedule: an open-label randomised controlled trial. Lancet Infect Dis. 2015 Feb;15(2):172-80. doi: 10.1016/S1473-3099(14)71057-6. Epub 2015 Jan 8. PMID 25577661
- [Derived] Khatami A, Clutterbuck EA, Thompson AJ, McKenna JA, Pace D, Birks J, Snape MD, Pollard AJ. Evaluation of the induction of immune memory following infant immunisation with serogroup C Neisseria meningitidis conjugate vaccines--exploratory analyses within a randomised controlled trial. PLoS One. 2014 Jul 14;9(7):e101672. doi: 10.1371/journal.pone.0101672. eCollection 2014. PMID 25020050